CLINICAL TRIAL: NCT00688441
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Nasal Carbon Dioxide in the Treatment of Seasonal Allergic Rhinitis
Brief Title: The Effect of Nasal Carbon Dioxide (CO2) in the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Kristen Yen, Associate Director, Clinical, Capnia, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C215
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Randomized; Double-Blind; Multi-Center; Placebo-Controlled; Phase II; Nasal Carbon Dioxide; Carbon Dioxide; Efficacy; Safety; Total Nasal Symptom Score; RQLQ
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): CO2 Gas
  Interventions: Drug: Nasal CO2
- Placebo (Placebo Comparator): Inactive Placebo Gas
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nasal CO2 — Twice daily during the 14 day Treatment Period
  Arms: Active
Drug: Placebo — Use of the study drug dispenser at the same frequency as the active arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effect of nasal carbon dioxide in the treatment of Seasonal Allergic Rhinitis

DETAILED DESCRIPTION:
This multi-center, randomized, double-blind, placebo-controlled, parallel group trial will evaluate the efficacy and safety of a nasal, non-inhaled administration of carbon dioxide (CO2) in patients with seasonal allergic rhinitis. An estimated 500 patients who meet the eligibility criteria will be enrolled into this study at approximately 25 sites to ensure that approximately 400 patients are randomized and complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand informed consent and voluntarily consent to sign the informed consent form
* Able to comply with the requirements of the protocol (e.g., complete the diary within the protocol-specified window)
* Minimal 2-year history of Fall seasonal allergic rhinitis requiring pharmacotherapy
* Positive skin test to one or more Fall seasonal allergen (e.g., ragweed, birch pollen, etc.)
* Females of childbearing potential must commit to using an acceptable method of birth control and have a negative pregnancy test

Exclusion Criteria:

* History of asthma (other than mild intermittent)
* Acute or significant sinusitis or upper respiratory infection within 14 days of enrollment
* Existing serious medical condition (e.g., severe emphysema) that precludes participation
* Females who are pregnant or breast-feeding and/or who plan to become pregnant or to breast-feed during the study participation or within 7 days after the last study drug administration
* Initiation of immunotherapy or have a change in immunotherapy dose within the 6 months preceding enrollment (if on immunotherapy, the same dose must be maintained throughout the trial)
* Planned travel outside the study area for the duration of study period
* Participation in another clinical study within 30 days of planned enrollment date and for the duration of the study
* Participation in a previous study with Nasal CO2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The mean change in reflective Total Nasal Symptom Score (TNSS) over the Treatment Period compared to baseline in nasal CO2 or placebo | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: S. David Miller, MD, Study Chair — Northeast Medical Research Associates, Inc.